CLINICAL TRIAL: NCT04768751
Title: Assessment of Acute Kidney Injury as a Risk Factor for Myocardial Injury and Ventricular Systolic Dysfunction After Non-Cardiac Surgery in Critical Patients
Brief Title: Acute Kidney Injury as a Risk Factor for Myocardial Injury and Ventricular Dysfunction
Status: Completed | Type: Observational
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Alaa Ali M. Elzohry, 4- Lecturer of Anesthesia, ICU and Pain Relief, South Egypt Cancer Institute, Assiut University, Egypt, South Egypt Cancer Institute
Other Study IDs: Acute Kidney injury
Record Dates: First submitted 2021-02-20; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Acute Kidney Injury; Ventricular Dysfunction; Myocardium; Injury
MeSH Terms: conditions — Acute Kidney Injury; Ventricular Dysfunction; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: kidney assessment — Urea, BUN, and Creatinine BLOOD LEVELS

SUMMARY:
Acute kidney injury (AKI) is classically described as an abrupt or rapidly reversible reduction in the excretion of nitrogenous waste products, including urea, nitrogen and creatinine. Acute kidney injury definition emphasizes on the filtration function of the kidney, a measure that is unique and easily and routinely measured .

Acute kidney injury is associated with significantly increased resource utilization and health care costs.

Major adverse cardiac events (MACE) after non cardiac surgery are a leading cause of morbidity and mortality. The reported incidence of postoperative myocardial infarction (POMI) among patients undergoing non cardiac surgery is between 3% and 6%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal kidney functions and free normal heart functions, were enrolled to this study

Exclusion Criteria:

* patients with chronic kidney disease, cardiac disease, who with minor operations, or emergency, were excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with normal kidney functions and free normal heart functions
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
development myocardial injury | through study completion, an average of 15 days
  New echocardiographic findings suggestive of ischemia (new regional wall motion abnormalities) or cardiac troponin T >.0.32 ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Alaa Ali Elzohry, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided